CLINICAL TRIAL: NCT01388127
Title: Minocycline Treatment in Acute Hemorrhagic Stroke for Evaluation of Treatment Efficacy and Blood Brain Barrier Permeability
Brief Title: Minocycline Treatment in Acute Hemorrhagic Stroke
Acronym: Minocycline
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Wolfson Medical Center (Other Government)
Responsible Party: Yair Lampl MD, Wolfson Medical Center
Other Study IDs: 0048-11 WOMC
Record Dates: First submitted 2011-07-03; First posted 2011-07-06 (Estimated); Last update posted 2011-07-06 (Estimated); Status verified 2011-06

CONDITIONS: Poor Performance Status

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The investigators will perform a double blind controlled study to investigate the efficacy of oral administration of 200 mg minocycline, on the neurological and functional outcome after acute hemorrhagic stroke and the effect on blood brain barrier permeability.

DETAILED DESCRIPTION:
Minocycline, a semisynthetic second generation derivative of tetracycline, was shown to have a clear beneficial neuroprotective effect in animal models of multiple sclerosis, Parkinson's disease, Huntington's disease and amyotrophic lateral sclerosis. Animal models provide promising evidence of minocycline's ability to improve outcomes in an animal stroke model.

In light of these findings, we will perform a double blind controlled study to investigate the efficacy of oral administration of 200 mg minocycline, on the neurological and functional outcome after acute hemorrhagic stroke and the effect on blood brain barrier permeability.

ELIGIBILITY:
Inclusion Criteria:

* Patients with acute hemorrhagic stroke

  1. age > 18
  2. NIHSS score > 5
  3. onset of stroke 6 to 24 hours prior to beginning of treatment. Patients, who arrived within 0 to 6 hours post stroke, were treated with other medications according to the best accepted medical treatment guidelines.

Exclusion Criteria:

1. Evidence of other disease of the central nervous system, including brain tumor, demyelinating disease, inflammatory disease of the central nervous system, craniotomy in the past, severe brain injuries and benign intracranial hypertension
2. pre-existing neurological disability
3. known allergic response to tetracyclines
4. acute or chronic renal failure
5. pre-existing infectious disease requiring antibiotic therapy
6. swallowing difficulties

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 150 patients after acute hemorrhagic stroke. Half treated with Minocycline.
Sampling Method: Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2011-07; Primary Completion 2012-07 (Estimated); Study Completion 2012-07 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Yair Lampl, MD, Principal Investigator — Edith Wolfson Medical Center
Locations (1):
- Edith Wolfson Medical Center, Holon, Israel, Israel